CLINICAL TRIAL: NCT01261013
Title: Intrastromal Corneal Ring Segment Implantation in 219 Keratoconic Eyes at Different Stages
Status: Completed | Type: Observational
Sponsor: Fernandez-Vega Ophthalmological Institute (Other)
Other Study IDs: IOFV-1
Record Dates: First submitted 2010-12-14; First posted 2010-12-16 (Estimated); Last update posted 2010-12-27 (Estimated); Status verified 2010-11

CONDITIONS: Keratoconus
Keywords: Keratoconus; intrastromal corneal ring segment; To evaluate the visual and refractive outcomes of intrastromal corneal ring segment in keratoconic eyes at different stages
MeSH Terms: conditions — Keratoconus

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- keratoconus stage I in whom KeraRing ICRS were implanted
- keratoconus stage II in whom KeraRing ICRS were implanted
- keratoconus stage III in whom KeraRing ICRS were implanted

SUMMARY:
The purpose of this study is to properly analyse the visual and refractive outcomes of implantation of KeraRing intrastromal corneal ring segment (ICRS) at the different stages of keratoconus.

ELIGIBILITY:
Inclusion Criteria:

* Patients who had keratoconus
* Contact lens intolerance and clear cornea.
* The maximum keratometric reading was less than 60.00 diopters (D)
* The minimum corneal thickness more than 300 μm.

Exclusion Criteria:

* Acute or grade IV keratoconus.
* Previous corneal or intraocular surgery.
* Cataract, history of glaucoma or retinal detachment, macular degeneration or retinopathy, neuro-ophthalmic diseases, and history of ocular inflammation

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients with keratoconus (stage I; stage II and stage III,according to the Amsler-Krumeich keratoconus classification) in whom KeraRing ICRS were implanted at the Fernández-Vega Ophthalmological Institute, Oviedo, Spain.
Sampling Method: Non-Probability Sample
Enrollment: 219 (Actual)
Dates: Start 2008-01; Study Completion 2010-03